CLINICAL TRIAL: NCT01697397
Title: A Feasibility Study For Monitoring And Recording Gastrointestinal Myoelectric Activity In Subjects With Suspected Or Diagnosed Irritable Bowel Syndrome (IBS) And Reports Of GI Pain And Asymptomatic Subjects Without IBS and GI Pain
Brief Title: Gastrointestinal Myoelectric Activity Protocol, the G-Tech EEnG Protocol
Status: Completed | Type: Observational
Sponsor: G-Tech Corporation (Industry)
Collaborators: Eminence Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-2012-001
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2024-01-23 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Gastrointestinal Diseases
Keywords: Irritable bowel syndrome; IBS; Gastrointestinal pain; Gastrointestinal functional disorder
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with and without FGIDs/IBS: Patients with functional gastro-intestinal disorders (FGIDs) undergo recording of myoelectric signals before, during, and after a meal. In addition, patients without FGIDs undergo recording of myoelectric signals before, during, and after a meal.
  Interventions: Device: Recording of Myoelectric Signals

INTERVENTIONS:
Device: Recording of Myoelectric Signals — Obtain recordings of the electrical signals of the gut.

SUMMARY:
A feasibility study for monitoring and recording gastrointestinal (GI) myoelectric activity in subjects with suspected or diagnosed irritable bowel syndrome (IBS) and reports of GI pain and asymptomatic subjects without IBS and GI pain.

DETAILED DESCRIPTION:
This single arm, prospectively enrolling, non-randomized feasibility study has been designed to transcutaneously detect and monitor myoelectric intestinal signals temporally associated with the symptoms of patients who report pain and have suspected or diagnosed IBS, and in controls [subjects without suspected IBS or diagnosis of IBS and prior and/or current complaints of pain].

ELIGIBILITY:
General Eligibility Criteria:

General Inclusion Criteria

* Willing and able to provide informed consent;
* Eighteen (18) years of age or older;
* Willing and able to follow a specified study procedure regimen;
* No known allergy to commercially available food or drink required by specified study procedure regimen;
* Willing and able to recline and remain still during the recordings.

General Exclusion Criteria

* Subject has an implantable device such as a pacemaker, defibrillator, nerve stimulator, insulin pump, automatic analgesic pump, or other automated implanted medical device;
* Known allergy to isopropyl (rubbing) alcohol;
* Known allergy to Ag/AgCl electrodes;
* Known allergy to glue adhesive (electrode adhesive);
* Dietary restrictions not permitting intake of food or drink required by this protocol;
* Dietary restrictions not permitting four (4) hour fasting period prior to start of myoelectric recording;
* Subject is pregnant or suspects pregnancy;
* Open sores or wounds on the abdomen;
* Any injury in or around the area of electrode placement that would cause pain with gentle pressure required for electrode and lead wire placement;
* Weight > 300 lbs (136 Kg) (excess weight can interfere with quality of the signals).

IBS With Complaints of GI Pain Eligibility Criteria IBS With Complaints of Pain Inclusion Criteria All answers must be "YES" to the All of the Following Inclusion Criteria Prior diagnosis of IBS and complaints of GI pain IBS With Complaints of Pain Exclusion Criteria All answers must be "NO" to the All of the Following Exclusion Criteria Functional dyspepsia; No reports of GI pain, past or present.

Control Subjects Eligibility Criteria Subjects who do NOT have a prior diagnosis of functional GI disorder

Control Subjects Inclusion Criteria All answers must be "YES" to the All of the Following Inclusion Criteria

No prior diagnosis IBS; No complaints of GI pain.

Control Subjects Exclusion Criteria All answers must be "NO" to the All of the Following Exclusion Criteria Current diagnosis of any GI disorder; Current or recent complaints of GI pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Irritable bowel syndrome, functional bowel disorder.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2012-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prince Shah, MD, Study Chair — G-Tech Chief Medical Officer and Medical Monitor
Locations (1):
- G-Tech Corporation, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Present in abstracts at society meetings and enter on-line on this website.

REFERENCES:
- [Result] Triadafilopoulos, George, et al.

RESULTS

PARTICIPANT FLOW:
Groups:
- Investigational Device Arm: 88 individuals were studied. Of the 88 individuals, 77 with FGID symptoms (constipation, diarrhea, pain, bloating) and 11 nominally healthy controls were studied. Data from the subjects were normalized to allow quantitative comparisons. Peaks in the frequency spectrum presumably due to motor activity were algorithmically identified and their total volume calculated. This was performed for the pre-prandial hour, a post-prandial 40-minute period and the final hour.
Period: Overall Study
Arm/Group | Investigational Device Arm
Started | 88
Completed | 88
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All 88 individuals met the eligibility criteria as described in the previous section and received the investigational device
Groups:
- Investigational Device Arm: 88 individuals participated in this study. Data from all the subjects were normalized to allow quantitative comparisons. Peaks in the frequency spectrum presumably due to motor activity were algorithmically identified and their total volume calculated. This was performed for the pre-prandial hour, a post-prandial 40-minute period and the final hour.
Arm/Group | Investigational Device Arm
Number analyzed (Participants) | 88
Age, Continuous [Mean (Full Range); unit: years] | 48.9 [22.0 to 81.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 31
Race/Ethnicity, Customized [Number; unit: participants]
  Race - Asian | 6
  Race - Caucasian | 68
  Race - Hispanic or Latino | 14
Region of Enrollment [Number; unit: participants]
  United States | 88
Number of Participants with FGID symptoms and those who denied having FGID symptoms [Count of Participants; unit: Participants]
  FGID Symptoms present | 77
  FGID symptoms absent (healthy controls) | 11

OUTCOME MEASURES:

1. Primary Outcome: Device Success Defined as the Ability to Record Myoelectric Signals in Study Subjects.
Description: All patients in the study received the investigational device for recording myoelectric signals. Patients had a variety of symptoms and diagnoses, among which the mean peak volume profiles for a group of subjects with gastroparesis (7 tests) and reflux disorder (9 tests) were identified and analyzed separately. Subjects were fed a 700 kCal meal 60 minutes into the test. Time-dependent peaks in the frequency spectra were identified and volumes (height x width x duration) were calculated from data obtained in 101 tests of FGID patients and controls. Peaks were associated with each of the digestive organs in frequency ranges as follows for stomach: 2-4 cycles per min. (cpm); small intestine: 5-12 cpm; and colon: 12-25 cpm. The patches measure the myoelectric voltage present at the skin surface to determine the motor activity of each organ. The unit of measure for the activity is (mV)**2 X Hz. This is a standard measurement used in frequency spectrum analysis.
Time Frame: Up to 4 hours at time of procedure
Measure: Number; unit: participants
Groups:
- Investigational Device Arm: 88 individuals in all were studied. 77 individuals reported having FGID symptoms (constipation, diarrhea, pain, bloating) and 11 individuals denied having any FGID symptoms. Data from all subjects were normalized to allow quantitative comparisons. Peaks in the frequency spectrum linked to gastrointestinal motor activity were algorithmically identified and their total volume calculated. This was performed for the pre-prandial hour, a post-prandial 40-minute period and the final hour.
Arm/Group | Investigational Device Arm
Number analyzed (Participants) | 88
participants | 88

2. Secondary Outcome: Secondary Efficacy Outcome
Description: The study was not powered to analyze the differences for the FGID conditions of constipation and diarrhea, but was for a group of subjects with gastroparesis and reflux disorder. For these two groups, the mean myoelectrical activity in the stomach, small intestine, and colon were calculated and compared to that of the health controls.
Time Frame: Up to 4 hours at time of procedure
Population: Among the subjects studied, a sub group of subjects reported having gastroparesis and reflux disorders. These subjects were analyzed as separate groups and compared to the subjects who denied having any gastrointestinal disorders.
Measure: Mean (Standard Deviation); unit: (mV)^2 x Hz
Groups:
- Individuals Without FGID Symptoms (Healthy Controls): 11 individuals who denied FGID symptoms served as healthy controls
- Individuals With Gastroparesis: Among the subjects with FGIDs, there were 7 tests conducted with individuals diagnosed with gastroparesis.
- Individuals With Reflux Disorder: 9 individuals were studied having been diagnosed with a reflux disorder
- Individuals With Bloating: 12 Individuals studied were diagnosed with bloating.
- Individuals With Constipation: 30 individuals studied were diagnosed with constipation.
- Individuals With Diarrhea: 18 individuals studies were diagnosed with diarrhea.
Arm/Group | Individuals Without FGID Symptoms (Healthy Controls) | Individuals With Gastroparesis | Individuals With Reflux Disorder | Individuals With Bloating | Individuals With Constipation | Individuals With Diarrhea
Number analyzed (Participants) | 11 | 7 | 10 | 12 | 30 | 18
(mV)^2 x Hz
  Stomach Preprandial myoelectrical activity | 2.14 (1.27) | 0.75 (0.82) | 0.78 (0.61) | 1.24 (1.56) | 1.89 (1.88) | 1.61 (1.62)
  Stomach Postprandial myoelectrical activity 1st hr | 4.75 (2.82) | 1.54 (0.86) | 5.16 (4.90) | 5.02 (5.68) | 8.62 (15.67) | 3.53 (2.79)
  Stomach Postprandial myoelectrical activity 2nd hr | 7.39 (8.00) | 1.57 (0.87) | 11.41 (20.70) | 9.29 (17.40) | 7.19 (5.75) | 3.91 (3.06)
  Intestine Preprandial myoelectrical activity | 16.27 (15.16) | 7.68 (6.09) | 10.24 (8.67) | 12.04 (9.39) | 11.49 (6.72) | 14.55 (9.94)
  Intestine Postprandial myoelectrical activity 1st hr | 24.46 (11.55) | 9.38 (5.94) | 16.36 (8.78) | 24.01 (15.06) | 16.87 (8.11) | 21.79 (14.80)
  Intestine Postprandial myoelectrical activity 2nd hr | 20.18 (10.49) | 10.03 (8.54) | 15.28 (6.88) | 20.76 (11.42) | 14.33 (7.42) | 19.17 (15.49)
  Colon Preprandial myoelectrical activity | 3.32 (3.81) | 4.39 (4.05) | 8.60 (14.54) | 9.24 (11.91) | 7.50 (8.98) | 6.43 (7.25)
  Colon Postprandial myoelectrical activity 1st hr | 5.25 (2.42) | 11.83 (12.43) | 3.98 (4.02) | 4.49 (2.76) | 5.01 (6.24) | 10.68 (13.78)
  Colon Postprandial myoelectrical activity 2nd hr | 7.24 (4.26) | 9.26 (6.60) | 3.81 (2.80) | 8.20 (4.84) | 8.28 (9.28) | 7.39 (9.07)

3. Secondary Outcome: Number of Anticipated, Un-Anticipated, and Serious Adverse Events
Description: Assess and record anticipated adverse events (AEs), unanticipated adverse device effects (UADEs), and serious adverse events (SAEs) at time of recording
Time Frame: Up to 4 hours at time of procedure
Measure: Number; unit: adverse events
Groups:
- Investigational Device Arm: 77 individuals with FGID's and 11 individuals without FGID's were studied.
Arm/Group | Investigational Device Arm
Number analyzed (Participants) | 88
adverse events | 0

ADVERSE EVENTS:
Groups:
- Investigational Device Arm: 77 patients with FGID symptoms (constipation, diarrhea, pain, bloating) and 11 nominally healthy controls were tested. Data from different subjects were normalized to allow quantitative comparisons. Peaks in the frequency spectrum presumably due to motor activity were algorithmically identified and their total volume calculated. This was performed for the pre-prandial hour, a post-prandial 40-minute period and the final hour.
Arm/Group | Investigational Device Arm
Serious Adverse Events (participants affected / at risk) | 0/88
Other Adverse Events (participants affected / at risk) | 0/88

LIMITATIONS AND CAVEATS:
This 3 hour clinical trial was carried out as an investigation to determine the viability of a wireless, waterproof patch based system. 3 days of data would provide full coverage of all GI events, and nearly 5x the statistical precision of this test.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No